CLINICAL TRIAL: NCT04923438
Title: The Effect of Telerehabilitation on the Quality of Life, Anxiety and Depression Levels of Children With Cerebral Palsy and Their Caregivers
Brief Title: The Effect of Telerehabilitation on the Children With Cerebral Palsy and Their Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2021.180
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; telerehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telerehabilitation (Experimental): The exercises will be applied twice a week for a total of 12 weeks, and each program will last roughly 30 minutes.
  Interventions: Other: Telerehabilitation
- control (Active Comparator): The same exercise program will be prepared and given as a printout and they will be asked to do their exercises at home. This group will also be included in the study as a control group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Telerehabilitation — The exercise program will begin with a warm-up, followed by a stretching exercise and an alphabetical exercise game called what's your name, and will end with a cool-down. The exercises will be performed 2 times a week for a total of 12 weeks, and each program will last for roughly 30 minutes. it will last. In what is your name game, 10 5-letter words containing the whole alphabet were produced and children will work out the exercises corresponding to each letter with a word they choose for each day.
  Arms: telerehabilitation
Other: Control — The same exercise program will be prepared and given to the patients who are offered and not accepted telerehabilitation, and they will be asked to do their own exercises at home. This group will also be included in the study as a control group.
  Arms: control

SUMMARY:
Cerebral palsy develops due to brain damage before, during and after birth. Motor control is impaired in individuals with cerebral palsy. Disturbances occur in muscle tone, mobility and body posture. There is no definitive treatment for cerebral palsy, but improvement in functions can be achieved with physiotherapy.

Because of the covid-19 pandemic precautions, activity level has been decreasing in children with cerebral palsy, as in adults.

Children experience physical, social and psychological problems caused by physical inactivity.

Exercises and games that can be done comfortably in the house will positively affect the physical development of children and enable them to spend productive time by getting away from excessive technology, internet and smart phone usage, excessive screen time.

The aim of this project; To ensure that children with cerebral palsy who need intense exercise and activity and who experience physical inactivity due to COVID-19 can exercise with telerehabilitation and to determine the effect of telerehabilitation on the quality of life, anxiety and depression levels of children with cerebral palsy and their caregivers.

It will be compared to a control group that did not accept telerehabilitation but was recommended to exercise at home.

DETAILED DESCRIPTION:
Cerebral palsy (SP); It is a group of permanent neuromotor disorders affecting movement, muscle tone and posture development as a result of non-progressive damage to the brain in the prenatal and neonatal period. In children with CP, it is observed that primitive reflexes continue, correction reactions occur late, muscle weakness, spasticity, loss of coordination and normal motor control cannot develop. Clinically SP; Spastic, dyskinetic, ataxic and mixed types are divided into four groups as SP.

Although there is no definitive treatment for CP, physiotherapy applications are of great importance in the treatment of problems. With physical therapy exercises, it is known that children with CP progress in factors such as postural control, muscle strength, flexibility, balance, physical activity capacity, mental well-being, participation in social life.

The COVID-19 (coronavirus) pandemic, which has recently surrounded the whole world, has caused serious measures to be taken in all areas in our country. Serious warnings are made that everyone should stay at home. During this period, physical activity levels of children as well as adults decreased significantly. Children experience physical, social and psychological problems caused by physical inactivity.

Exercises and games that can be done easily in the house will positively affect the physical development of children and enable them to spend productive time by getting away from excessive technology, internet and smart phone usage, excessive screen time. (aerobic) and stretching activities. Physical activity programs that are age-appropriate, fun and diverse should be created for children.

In addition, games for physical activity in the family; It is also thought that it will increase socialization within the family, that individuals will listen to each other more, understand, share more, and prevent some anxiety and stress caused by coronavirus.

The aim of this project; To ensure that children with cerebral palsy who need intense exercise and activity and who experience physical inactivity due to COVID-19 can exercise with telerehabilitation and to determine the effect of telerehabilitation on the quality of life, anxiety and depression levels of children with cerebral palsy and their caregivers. It will be compared to a control group that did not accept telerehabilitation but was recommended to exercise at home.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Spastic Hemiplegic and Diplegic Cerebral Palsy in participating children confirmed by pediatric neurologists

Being GMFCS I and II

Spasticity value of 1, 2 or maximum 3 in the evaluation made with Modified Ashworth Scale (MAS) on lower extremity muscles

Being able to stand and walk without using any auxiliary equipment

Being mentally capable of reading the commands of the assessment.

Agree to participate in the study

Exclusion Criteria:

Not having ambulation

Having a cognitive disorder

Having undergone any orthopedic surgery or spasticity replacement procedure in the past 12 months

Having vision problems except refraction

Having any known systemic problems

Having an uncontrolled epileptic seizure

Having lower extremity contracture that affects the evaluation

The occurrence of any health problems that could affect the work

Refusing to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-06-12 (Estimated); Study Completion 2021-06-26 (Estimated)

PRIMARY OUTCOMES:
CP-QOL-Child ve Teen | Day 0 - Day 90
  Evaluates the quality of life in Cerebral Palsy.
Revised Child Anxiety and Depression Scale | Day 0 - Day 90
  It was developed to screen for anxiety disorders and depression.
STAI-State Trait Anxiety Inventory | Day 0 - Day 90
  It is a self-evaluation questionnaire consisting of short statements.
BECK Depression Inventory | Day 0 - Day 90
  It will be applied in determining depression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag-Saygi, Prof. Dr., Study Chair — Physical Medicine and Rehabilitation Department, School of Medicine, Marmara University, Istanbul; Ayca Evkaya Acar, Lecturer, Principal Investigator — Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istanbul Medeniyet University; Nurahsen Demir, Res. Asst., Principal Investigator — Physical Medicine and Rehabilitation Department, School of Medicine, Marmara University, Istanbul
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Berker AN, Yalcin MS. Cerebral palsy: orthopedic aspects and rehabilitation. Pediatr Clin North Am. 2008 Oct;55(5):1209-25, ix. doi: 10.1016/j.pcl.2008.07.011. PMID 18929061
- [Background] Tilton AH. Management of spasticity in children with cerebral palsy. Semin Pediatr Neurol. 2004 Mar;11(1):58-65. doi: 10.1016/j.spen.2004.01.008. PMID 15132254
- [Background] Patel DR, Neelakantan M, Pandher K, Merrick J. Cerebral palsy in children: a clinical overview. Transl Pediatr. 2020 Feb;9(Suppl 1):S125-S135. doi: 10.21037/tp.2020.01.01. PMID 32206590
- [Background] McBurney H, Taylor NF, Dodd KJ, Graham HK. A qualitative analysis of the benefits of strength training for young people with cerebral palsy. Dev Med Child Neurol. 2003 Oct;45(10):658-63. doi: 10.1017/s0012162203001233. PMID 14515936